CLINICAL TRIAL: NCT00198029
Title: An Open Label Trial for Treating Carpometacarpal Osteoarthritis of the Thumb: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Genzyme, a Sanofi Company (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23034; 101584; Grant# K23AR050607-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2013-06-10 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Carpometacarpal Osteoarthritis
Keywords: Osteoarthritis; Hyaluronan; Carpometacarpal; Outcomes
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pilot Study of Hylan G-F 20 (Experimental): 32 Subjects have received Synvisc Injections and followed for 6 months.
  Interventions: Device: Synvisc (hylan G-F20)

INTERVENTIONS:
Device: Synvisc (hylan G-F20) — 32 subjects in the pilot study have received 3 1ml injections of Synvisc intraarticular over the course of 3 weeks and then followed for 6 months post injection

SUMMARY:
The purpose of this study is to find out if hyaluronan, an injectable medication for knee arthritis, also works for arthritis at the base of the thumb. This study will also evaluate how good ultrasound is at visualizing medication in the thumb joint. We are no longer recruiting for this part of the open label trial.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic evidence of at least moderate narrowing (joint space < 1mm) or the presence of osteophytes or sclerosis at the Carpometacarpal joint
* Patient complaint of unacceptable pain despite modification of activity, a trial of splinting and a therapeutic dose of NSAIDS
* If bilateral disease, only the most severely involved hand, (as defined by VAS for pain), will be entered in the study.
* Proficiency in English.

Exclusion Criteria:

* Previous bad injury to the thumb
* Previous hand surgery on the study thumb
* Known hand comorbidities (i.e. carpal tunnel syndrome, de Quervains Tenosynovitis etc)
* Rheumatoid arthritis or lupus
* Bleeding problems
* Being on blood thinners (except aspirin)
* Known allergies to any of the medications being used
* Allergies to chicken products
* Current use of oral steroids
* Cancer that is not cured or in remission
* Severe diabetes
* A serious infection somewhere else in the subject's body

Ages: 45 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Mandl, MD MPH, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Derived] Mandl LA, Hotchkiss RN, Adler RS, Lyman S, Daluiski A, Wolfe SW, Katz JN. Injectable hyaluronan for the treatment of carpometacarpal osteoarthritis: open label pilot trial. Curr Med Res Opin. 2009 Sep;25(9):2103-8. doi: 10.1185/03007990903084016. PMID 19601706

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with painful CMC OA and radiographic changes of Kellgren and Lawrence (K+L) Grade 2-4 were recruited from rheumatology and hand surgery practices at the Hospital for Special Surgery from 2004-2005
Pre-assignment Details: Exclusion criteria included: age < 45, systemic rheumatic disease, self-reported comorbid hand conditions, history of gout or pseudogout, bleeding diatheses, previous surgery to the involved thumb, and no evidence of CMC joint space narrowing. Patients must have failed some form of conservative therapy, such as NSAIDS, acetaminophen or splinting.
Groups:
- Synvisc Group: Thirty-two patients were injected once weekly for three weeks with Hylan G-F 20 and followed for 6 months post injections.
Period: Overall Study
Arm/Group | Synvisc Group
Started | 32
Completed | 28
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: The average baseline VAS for pain was 62(range 38-100), and DASH was 29.7 (range 1- 68). 53% had ≥ 1 previous corticosteroid injection. All patients had moderate or severe radiographic OA of the CMC joint: 59% were K+L Grade 4, 25% Grade 3, and 16% Grade 2. No patients had clinical evidence of carpal tunnel syndrome or DeQuervain's tenosynovitis.
Groups:
- Open Label Group: Thirty-two patients were injected over ten months with Synvisc and followed for 6 months post injections.
Arm/Group | Open Label Group
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: The Disabilities of the Arm, Shoulder and Hand Outcome Measure
Description: The DASH Outcome Measure is a 30-item, self-report questionnaire designed to measure physical function and symptoms in people with any of several musculoskeletal disorders of the upper limb. Scores are transformed to a 0-100 scale, with a higher value indicating greater disability. The change in DASH (delta) over those 6 months was recorded.
Time Frame: 26 weeks (6 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synvisc Group
Number analyzed (Participants) | 32
units on a scale | 12.6 (17.2)

2. Secondary Outcome: Visual Analog Scale for Pain
Description: The visual analog scale for pain (VAS) is a test requiring a patient to indicate along a line how much pain they are experiencing between 0-100. A score of 100 indicates the maximum possible pain level and a score of 0 indicates no pain. Scores are recorded as whole number integers. The change in VAS (delta) over those 6 months was recorded.
Time Frame: 26 weeks (6 months)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Synvisc Group
Number analyzed (Participants) | 32
mm | 15.2 (29.5)

ADVERSE EVENTS:
Arm/Group | Open Label Group
Serious Adverse Events (participants affected / at risk) | 3/32
Other Adverse Events (participants affected / at risk) | 3/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Group (N=32)
Unlikely Related Pseudogout (Musculoskeletal and connective tissue disorders) | 1 (1) — One patient had an acute attack of crystal proven pseudogout in the ipsilateral wrist 33 days after the last CMC hyaluronic acid injection. The patient had no previous history of inflammatory arthritis and had been well in the interim.
Unlikely Related GI Bleed (Gastrointestinal disorders) | 1 (1) — A 74 year old patient withdrew after a gastrointestinal bleed that occurred 69 days after the last HA injection.
Possibly but Unlikely Related Fall (Musculoskeletal and connective tissue disorders) | 1 (1) — One patient slipped on the way to the hospital for the third HA injection and suffered a broken scapula; this patient completed the study.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Group (N=32)
Pain at Injection Site (Musculoskeletal and connective tissue disorders) | 3 (96) — Out of the 96 total injections, 3 resulted in post-injection pain and swelling requiring treatment. Two were after the second injection, and one was after the third injection. All symptoms rapidly resolved with ice, NSAIDS or COX-2 inhibitor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No